CLINICAL TRIAL: NCT00136864
Title: The Impact of Positron Emission Tomography (PET) Imaging in Stage III Non-small Cell Lung Cancer: A Prospective Randomized Clinical Trial (PET START Trial)
Brief Title: Positron Emission Tomography (PET) Imaging in Stage III Non-small Cell Lung Cancer (PET START Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTA-Control-087276
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Positron-Emission Tomography; PET Scan; Non-Small-Cell Lung Carcinoma; Diagnosis; Radiation Oncology; Lung Cancer; Randomized Controlled Trial; Oncology; Radiation Planning
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease; Lung Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PET Imaging
  Interventions: Procedure: PET Diagnostic Imaging
- 2 (No Intervention): Standard Imaging

INTERVENTIONS:
Procedure: PET Diagnostic Imaging — Patients in the PET group will undergo the standard diagnostic tests plus PET to determine those suitable for combined modality therapy
  Arms: 1

SUMMARY:
Locally advanced non-small cell lung cancer, NSCLC, (Stage III) is potentially curable with aggressive combined modality therapy (chemotherapy and radiation). Conventional imaging can only evaluate gross anatomic abnormalities but functional imaging with positron emission tomography (PET) may more accurately identify patients who will benefit from aggressive combined modality therapy.

This prospective randomized clinical trial will enroll 400 patients that have undergone conventional staging for lung cancer and have been found to have Stage III NSCLC. The patients will then be randomized to either standard combined modality therapy for Stage III NSCLC or to PET imaging prior to combined modality therapy with curative intent. Based on the PET findings, patients will either be suitable for combined modality therapy with curative intent or not.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of NSCLC. Must have documented pathology report with histology indicated (e.g. squamous, adenocarcinoma, large cell, NSCLC not otherwise specified).
* Stage III (mediastinal node positive) NSCLC based on conventional staging (e.g. computed tomography [CT] scan of chest and upper abdomen, CT or magnetic resonance imaging [MRI] of brain, bone scan).
* Suitable for combined modality (chemotherapy and radiation) therapy or radical radiation therapy or trimodality therapy (chemotherapy, radiation and surgery).

Exclusion Criteria:

* Stage IV NSCLC (by conventional staging).
* Small cell lung cancer.
* Poor performance status Eastern Cooperative Oncology Group (ECOG) 3-4.
* Poor pulmonary function precluding radical radiation therapy (Adequate pulmonary reserve for radical radiation therapy. Pulmonary function tests should have forced expiratory volume in 1 second (FEV1) > 1.0 liter or > 40% predicted, diffusing capacity of the lung for carbon monoxide (DLCO) > 45% and/or predicted contralateral FEV1 > 800 cc based on quantitative ventilation perfusion lung scan).
* Significant concurrent medical problems (e.g. uncontrolled diabetes, active cardiac problems, significant chronic obstructive pulmonary disease).
* Insulin dependent diabetic where requirements for PET imaging may be problematic.
* Unable to lie supine for at least 30 minutes in radiation treatment position for imaging with PET.
* Failure to provide informed consent.
* Previous PET scan relating to recent cancer diagnosis prior to entry into study.
* Pregnant or lactating females.
* Prior thoracic radiation.
* Prior malignancy within 3 years from randomization (except nonmelanotic skin cancer or carcinoma in situ of the cervix).
* Administered more than two cycles of chemotherapy prior to radical radiation therapy or concurrent chemoradiation (as part of induction or sequential chemotherapy prior to randomization) for the current malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2004-08; Primary Completion 2009-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Stage III NSCLC patients upstaged by PET | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Impact of PET on radiation treatment planning | 2 years
Prognostic ability of PET standard uptake value | 2 years
Number of patients downstaged by PET | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yee C Ung, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Mark N Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); William Evans, MD, Principal Investigator — Juravinski Cancer Centre
Locations (5):
- Canada (5):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Toronto-Sunnybrook Odette Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario